CLINICAL TRIAL: NCT01098110
Title: A Multicenter, Randomized, Double-blind, Fixed-dose, 6-week Trial of the Efficacy and Safety of Asenapine Compared With Placebo in Subjects With an Acute Exacerbation of Schizophrenia (Phase 3)
Brief Title: 6-week Trial of the Efficacy and Safety of Asenapine Compared to Placebo in Participants With an Acute Exacerbation of Schizophrenia (P06124)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P06124
Record Dates: First submitted 2010-04-01; First posted 2010-04-02 (Estimated); Results first posted 2015-04-17 (Estimated); Last update posted 2024-06-20 (Actual); Status verified 2022-02

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — asenapine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Asenapine 5 mg BID (Experimental): Participants received a 5 mg asenapine fast dissolving tablet twice daily (BID) for 6 weeks.
  Interventions: Drug: Asenapine 5 mg
- Asenapine 10 mg BID (Experimental): Participants received a 5 mg asenapine fast dissolving tablet BID on Day 1, then 10 mg asenapine fast dissolving tablet BID thereafter for a total of 6 weeks.
  Interventions: Drug: Asenapine 5 mg; Drug: Asenapine 10 mg
- Placebo BID (Placebo Comparator): Participants received matching placebo BID for 6 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Asenapine 5 mg — Asenapine 5 mg fast dissolving tablets sublingually without water twice daily, in the morning (around 8 am) and in the evening (around 8 pm), on Day 1 only or for 6 weeks.
  Other Names: SCH 900274
  Arms: Asenapine 10 mg BID; Asenapine 5 mg BID
Drug: Asenapine 10 mg — Participants receive on Day 2, 10 mg BID of fast dissolving tablets sublingually without water twice daily, in the morning (around 8 am) and in the evening (around 8 pm), for 6 weeks.
  Other Names: SCH 900274
  Arms: Asenapine 10 mg BID
Drug: Placebo — A matching placebo of asenapine sublingual tablet not containing asenapine
  Arms: Placebo BID

SUMMARY:
A multicenter, randomized, parallel-group, double-blind, fixed dose, 6-week trial of the efficacy and safety of asenapine compared with placebo in participants with an acute exacerbation of schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* current diagnosis of schizophrenia of paranoid, disorganized, catatonic, or undifferentiated (295.90) subtype
* minimum Positive and Negative Syndrome Scale (PANSS) total score of 60 at screening and Baseline.
* participant had a score of at least 4 in two or more of 5 items in the positive subscale of the PANSS at Screening and Baseline.
* participant confirmed by the investigator to be experiencing an acute exacerbation of schizophrenia as evidenced by ALL of the following:

  * at the screening test, the duration of the current episode was no more than 2 months;
  * current symptoms represented a dramatic and substantial change compared to the participant's symptomatic state prior to the emergence of the current episode;
  * participant was in need of changing medication or dosage to treat newly appeared or worsened positive symptoms.
* participant had a Clinical Global Impressions-Severity (CGI-S) scale score of at least 4 (moderately ill) at Baseline;
* responded positively to an antipsychotic medication in a prior episode.
* discontinued the use of all prohibited concomitant medications, with last dose taken no later than the evening prior to the baseline visit (For depot neuroleptic, discontinuation must have occurred more than 3 months prior to randomization).
* participants must agree to inpatient status for screening period and for up to 42 days of dosing and, for out-patient phase, had a caregiver or an identified responsible person (e.g., family member, social worker, case worker, or nurse) whom the investigator accepts and who has agreed to provide support to the participant to ensure compliance with study treatment, out-patient visits, and protocol procedures.

Exclusion Criteria:

* not be treatment-refractory defined by the following criteria: (1) had been treated with at least two different atypical anti-psychotic agents at dosages equivalent to or greater than 600 mg/day of chlorpromazine (12 mg /day of haloperidol) for more than 4 weeks, each without clinical response, or (2) has received clozapine for 12 weeks immediately preceding the screening.
* not have received treatment with 3 or more antipsychotic drugs, or dose-equivalents higher than 18 mg/day of haloperidol (equivalent 900 mg/day of chlorpromazine) within one month prior to randomization.
* not have a diagnosis of schizoaffective disorder; schizophrenia of residual subtype; schizophreniform disorder, or schizophrenia with course specifiers continuous, single episode in partial remission, or single episode in full remission
* not have a concurrent psychiatric disorder other than schizophrenia coded on Axis I; not have a primary diagnosis other than schizophrenia
* not have had a known diagnosis of borderline personality disorder, mental retardation or organic brain disorder.
* not have a 20% or greater decrease in PANSS total score from screening to baseline
* not have an imminent risk of self-harm or harm to others, in the investigator's opinion.
* not have a substance induced psychotic disorder or a behavioral disturbance thought to be due to substance abuse
* not be currently under involuntary in-patient confinement.
* not been previously treated with asenapine.

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 532 (Actual)
Dates: Start 2010-05-25 (Actual); Primary Completion 2014-04-14 (Actual); Study Completion 2014-04-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kinoshita T, Bai YM, Kim JH, Miyake M, Oshima N. Efficacy and safety of asenapine in Asian patients with an acute exacerbation of schizophrenia: a multicentre, randomized, double-blind, 6-week, placebo-controlled study. Psychopharmacology (Berl). 2016 Jul;233(14):2663-74. doi: 10.1007/s00213-016-4295-9. Epub 2016 Jun 8. PMID 27271087

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Asenapine 5 mg BID | Asenapine 10 mg BID | Placebo BID
Started | 176 (Randomized participants) | 182 (Randomized participants) | 174 (Randomized participants)
Treated | 175 (Received at least one dose of trial medication) | 181 (Received at least one dose of trial medication) | 174 (Received at least one dose of trial medication)
Completed | 114 | 109 | 80
Not Completed | 62 | 73 | 94
Not completed — Withdrawal by Subject | 14 | 24 | 19
Not completed — Adverse Event | 30 | 32 | 43
Not completed — Lack of Efficacy | 13 | 9 | 27
Not completed — Other | 4 | 7 | 5
Not completed — Untreated | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Participants who received at least one dose of trial medication.
Groups:
- Asenapine 5 mg BID: Participants received a 5 mg asenapine fast dissolving tablet BID for 6 weeks.
- Total: Total of all reporting groups
Arm/Group | Asenapine 5 mg BID | Asenapine 10 mg BID | Placebo BID | Total
Number analyzed (Participants) | 175 | 181 | 174 | 530
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.41 (11.00) | 41.72 (11.10) | 41.11 (12.27) | 41.42 (11.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100 | 82 | 93 | 275
  Male | 75 | 99 | 81 | 255

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Total Score.
Description: PANSS total score measures symptoms of schizophrenia and consists of responses to 30 items: 7 items from the positive subscale (P1-P7), 7 items from the negative subscale (N1-N7) and 16 items from the general psychopathology subscale (G1-G16). Responses to each item range from 1 = absence of symptom, to 7 = most extreme symptoms. The PANSS total score is the sum of the scores for all 30 items, and ranges from 30 to 210, with a higher score indicating greater severity of symptoms. Change from baseline values that are negative represent an improvement in symptoms.
Time Frame: Baseline and Day 42
Population: All randomized participants who received at least one dose of trial medication, and had baseline and at least one post-baseline PANSS measurement. Dropout or missing data are imputed by the last observation carried forward (LOCF) method.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Asenapine 5 mg BID | Asenapine 10 mg BID | Placebo BID
Number analyzed (Participants) | 173 | 178 | 174
Score on a scale | -12.24 [-15.28 to -9.20] | -14.17 [-17.12 to -11.22] | -0.95 [-3.95 to 2.06]
Statistical Analysis 1: Comparison: Asenapine 5 mg BID vs Placebo BID; Test type: Superiority or Other; p < 0.0001, ANCOVA — Statistical significant: p=<0.05, two sided; Change from baseline a response variable, baseline score a covariate, treatment groups and regions as explanatory variables; Least square (LS) means difference = -11.29, 95% CI 2-sided [-15.42 to -7.16], Standard Error of Mean 2.10 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 2: Comparison: Asenapine 10 mg BID vs Placebo BID; Test type: Superiority or Other; p < 0.0001, ANCOVA — Statistical significant: p=<0.05, two sided; [statistical method as in outcome 1, analysis 1]; LS mean difference = -13.22, 95% CI 2-sided [-17.33 to -9.12], Standard Error of Mean 2.09 — Asenapine 10 mg BID minus Placebo BID

2. Secondary Outcome: Change From Baseline in PANSS Positive Symptom Score.
Description: PANSS Positive subscale measures symptoms of schizophrenia and consists of responses to 7 items (P1-P7). Responses to each item range from 1 = absence of symptom, to 7 = most extreme symptoms. The PANSS Positive subscale sums all 7 items and ranges from 7 to 49, with a higher score indicating greater severity of symptoms. An improvement in symptoms is represented by change from baseline values that are negative.
Time Frame: Baseline and Day 42
Population: All randomized participants who received at least one dose of trial medication, and had baseline and at least one post-baseline PANSS measurement. Dropout or missing data are imputed by the LOCF method.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Asenapine 5 mg BID | Asenapine 10 mg BID | Placebo BID
Number analyzed (Participants) | 173 | 178 | 174
Score on a scale | -4.31 [-5.29 to -3.33] | -4.63 [-5.59 to -3.68] | -0.85 [-1.82 to 0.13]
Statistical Analysis 1: Comparison: Asenapine 5 mg BID vs Placebo BID; Test type: Superiority or Other; p < 0.0001, ANCOVA; Change from baseline a response variable, baseline score a covariate; Least square (LS) means difference = -3.47, 95% CI 2-sided [-4.80 to -2.13], Standard Error of Mean 0.68 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 2: Comparison: Asenapine 10 mg BID vs Placebo BID; Test type: Superiority or Other; p < 0.0001, ANCOVA; Change from baseline a response variable, baseline score a covariate; LS mean difference = -3.79, 95% CI 2-sided [-5.11 to -2.46], Standard Error of Mean 0.67 — Asenapine 10 mg BID minus Placebo BID

3. Secondary Outcome: Change From Baseline in PANSS Negative Symptom Score.
Description: PANSS Negative subscale measures symptoms of schizophrenia and consists of responses to 7 items (N1-N7). Responses to each item range from 1 = absence of symptom, to 7 = most extreme symptoms. The PANSS Negative subscale sums all 7 items and ranges from 7 to 49, with a higher score indicating greater severity of symptoms. . An improvement in symptoms is represented by change from baseline values that are negative.
Time Frame: Baseline and Day 42
Population: All randomized participants who received at least one dose of trial medication, and had baseline and at least one post-baseline PANSS measurement. One participant from the 5 mg BID arm was missing a post-baseline measurement. Dropout or missing data are imputed by the LOCF method.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Asenapine 5 mg BID | Asenapine 10 mg BID | Placebo BID
Number analyzed (Participants) | 172 | 178 | 174
Score on a scale | -2.72 [-3.50 to -1.93] | -3.27 [-4.03 to -2.51] | -0.24 [-1.02 to 0.53]
Statistical Analysis 1: Comparison: Asenapine 5 mg BID vs Placebo BID; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least square (LS) means difference = -2.47, 95% CI 2-sided [-3.53 to -1.41], Standard Error of Mean 0.54 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 2: Comparison: Asenapine 10 mg BID vs Placebo BID; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS mean difference = -3.03, 95% CI 2-sided [-4.08 to -1.97], Standard Error of Mean 0.54 — Asenapine 10 mg BID minus Placebo BID

4. Secondary Outcome: Change From Baseline in PANSS General Psychopathology Score.
Description: PANSS General Psychopathology subscale measures symptoms of schizophrenia and consists of responses to 16 items (G1-G16). Responses to each item range from 1 = absence of symptom, to 7 = most extreme symptoms. The PANSS General Psychopathology subscale is the sum of the scores for all 16 items and ranges from 16 to 112, with a higher score indicating greater severity of symptoms.. An improvement in symptoms is represented by change from baseline values that are negative.
Time Frame: Baseline and Day 42
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Asenapine 5 mg BID | Asenapine 10 mg BID | Placebo BID
Number analyzed (Participants) | 173 | 178 | 174
Score on a scale | -5.26 [-6.81 to -3.72] | -6.34 [-7.84 to -4.83] | 0.19 [-1.34 to 1.72]
Statistical Analysis 1: Comparison: Asenapine 5 mg BID vs Placebo BID; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least square (LS) means difference = -5.46, 95% CI 2-sided [-7.56 to -3.35], Standard Error of Mean 1.07 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 2: Comparison: Asenapine 10 mg BID vs Placebo BID; Test type: Superiority or Other; p < 0.0001, ANCOVA — Statistical significant: p=<0.05, two sided; [statistical method as in outcome 1, analysis 1]; LS mean difference = -6.53, 95% CI 2-sided [-8.62 to -4.44], Standard Error of Mean 1.06 — Asenapine 10 mg BID minus Placebo BID

5. Secondary Outcome: Change From Baseline in PANSS Marder Factor Positive Symptom Score.
Description: PANSS Marder Factor Positive symptom score measures symptoms of schizophrenia and consists of responses to 8 items (P1,P3,P5,P6,N7,G1,G9,G12). Responses to each item range from 1 = absence of symptom, to 7 = most extreme symptoms. The PANSS Marder Factor Positive symptom score is the sum of the scores for all 8 items and ranges from 8 to 56, with a higher score indicating greater severity of symptoms. An improvement in symptoms is represented by change from baseline values that are negative.
Time Frame: Baseline and Day 42
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Asenapine 5 mg BID | Asenapine 10 mg BID | Placebo BID
Number analyzed (Participants) | 173 | 178 | 174
Score on a scale | -4.78 [-5.75 to -3.81] | -5.03 [-5.98 to -4.09] | -1.37 [-2.33 to -0.41]
Statistical Analysis 1: Comparison: Asenapine 5 mg BID vs Placebo BID; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least square (LS) means difference = -3.41, 95% CI 2-sided [-4.72 to -2.09], Standard Error of Mean 0.67 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 2: Comparison: Asenapine 10 mg BID vs Placebo BID; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS mean difference = -3.66, 95% CI 2-sided [-4.97 to -2.35], Standard Error of Mean 0.67 — Asenapine 10 mg BID minus Placebo BID

6. Secondary Outcome: Change From Baseline in PANSS Marder Factor Negative Symptom Score.
Description: PANSS Marder Factor Negative symptom score measures symptoms of schizophrenia and consists of responses to 7 items (N1,N2,N3,N4,N6,G7,G16). Responses to each item range from 1 = absence of symptom, to 7 = most extreme symptoms. The PANSS Marder Factor Negative symptom score is the sum of the scores for all 7 items and ranges from 7 to 49, with a higher score indicating greater severity of symptoms. An improvement in symptoms is represented by change from baseline values that are negative.
Time Frame: Baseline and Day 42
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Asenapine 5 mg BID | Asenapine 10 mg BID | Placebo BID
Number analyzed (Participants) | 173 | 178 | 174
Score on a scale | -2.77 [-3.58 to -1.96] | -3.35 [-4.14 to -2.55] | -0.41 [-1.21 to 0.40]
Statistical Analysis 1: Comparison: Asenapine 5 mg BID vs Placebo BID; Test type: Superiority or Other; p < 0.0001, ANCOVA; Change from baseline a response variable, baseline score a covariate; Least square (LS) means difference = -2.36, 95% CI 2-sided [-3.47 to -1.26], Standard Error of Mean 0.56 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 2: Comparison: Asenapine 10 mg BID vs Placebo BID; Test type: Superiority or Other; p < 0.0001, ANCOVA; Change from baseline a response variable, baseline score a covariate; LS mean difference = -2.94, 95% CI 2-sided [-4.03 to -1.84], Standard Error of Mean 0.56 — Asenapine 10 mg BID minus Placebo BID

7. Secondary Outcome: Change From Baseline in PANSS Marder Factor Disorganized Thought Symptom Score.
Description: PANSS Marder Factor Disorganized Thought symptom score measures symptoms of schizophrenia and consists of responses to 7 items (P2,N5,G5,G10,G11,G13,G15). Responses to each item range from 1 = absence of symptom, to 7 = most extreme symptoms. The PANSS Marder Factor Disorganized Thought symptom score is the sum of the scores for all 7 items and ranges from 7 to 49, with a higher score indicating greater severity of symptoms. An improvement in symptoms is represented by change from baseline values that are negative.
Time Frame: Baseline and Day 42
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Asenapine 5 mg BID | Asenapine 10 mg BID | Placebo BID
Number analyzed (Participants) | 172 | 178 | 174
Score on a scale | -2.48 [-3.23 to -1.73] | -2.85 [-3.57 to -2.12] | 0.24 [-0.50 to 0.97]
Statistical Analysis 1: Comparison: Asenapine 5 mg BID vs Placebo BID; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least square (LS) means difference = -2.72, 95% CI 2-sided [-3.73 to -1.70], Standard Error of Mean 0.52 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 2: Comparison: Asenapine 10 mg BID vs Placebo BID; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS mean difference = -3.08, 95% CI 2-sided [-4.09 to -2.08], Standard Error of Mean 0.51 — Asenapine 10 mg BID minus Placebo BID

8. Secondary Outcome: Change From Baseline in PANSS Marder Factor Hostility/Excitement Symptom Score.
Description: PANSS Marder Factor Hostility/Excitement symptom score measures symptoms of schizophrenia and consists of responses to 4 items (P4,P7,G8,G14). Responses to each item range from 1 = absence of symptom, to 7 = most extreme symptoms. The PANSS Marder Factor Hostility/Excitement symptom score is the sum of the scores for all 4 items and ranges from 4 to 28, with a higher score indicating greater severity of symptoms. An improvement in symptoms is represented by change from baseline values that are negative.
Time Frame: Baseline and Day 42
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Asenapine 5 mg BID | Asenapine 10 mg BID | Placebo BID
Number analyzed (Participants) | 173 | 178 | 174
Score on a scale | -0.77 [-1.35 to -0.18] | -1.40 [-1.97 to -0.84] | 0.86 [0.28 to 1.43]
Statistical Analysis 1: Comparison: Asenapine 5 mg BID vs Placebo BID; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least square (LS) means difference = -1.62, 95% CI 2-sided [-2.41 to -0.83], Standard Error of Mean 0.40 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 2: Comparison: Asenapine 10 mg BID vs Placebo BID; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS mean difference = -2.26, 95% CI 2-sided [-3.04 to -1.47], Standard Error of Mean 0.40 — Asenapine 10 mg BID minus Placebo BID

9. Secondary Outcome: Change From Baseline in PANSS Marder Factor Anxiety/Depression Symptom Score.
Description: PANSS Marder Factor Anxiety/Depression symptom score measures symptoms of schizophrenia and consists of responses to 4 items (G2,G3,G4,G6). Responses to each item range from 1 = absence of symptom, to 7 = most extreme symptoms. The PANSS Marder Factor Anxiety/Depression symptom score is the sum of the scores for all 4 items and ranges from 4 to 28, with a higher score indicating greater severity of symptoms. An improvement in symptoms is represented by change from baseline values that are negative.
Time Frame: Baseline and Day 42
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Asenapine 5 mg BID | Asenapine 10 mg BID | Placebo BID
Number analyzed (Participants) | 173 | 178 | 174
Score on a scale | -1.55 [-2.01 to -1.08] | -1.67 [-2.12 to -1.22] | -0.13 [-0.59 to 0.32]
Statistical Analysis 1: Comparison: Asenapine 5 mg BID vs Placebo BID; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least square (LS) means difference = -1.41, 95% CI 2-sided [-2.04 to -0.78], Standard Error of Mean 0.32 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 2: Comparison: Asenapine 10 mg BID vs Placebo BID; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS mean difference = -1.53, 95% CI 2-sided [-2.16 to -0.91], Standard Error of Mean 0.32 — Asenapine 10 mg BID minus Placebo BID

10. Secondary Outcome: Percentage of Participants Who Were PANSS Responders.
Description: PANSS total score measures symptoms of schizophrenia and consists of responses to 30 items: 7 items from the positive subscale (P1-P7), 7 items from the negative subscale (N1-N7) and 16 items from the general psychopathology subscale (G1-G16). Responses to each item range from 1 = absence of symptom, to 7 = most extreme symptoms. The PANSS total score is the sum of the scores for all 30 items, and ranges from 30 to 210, with a higher score indicating greater severity of symptoms. The PANSS total score was determined at baseline and then at Day 42, and a participant with a 30% or greater reduction from baseline in PANSS total score at Day 42 was considered a PANSS responder.
Time Frame: Day 42
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Asenapine 5 mg BID | Asenapine 10 mg BID | Placebo BID
Number analyzed (Participants) | 173 | 178 | 174
Percentage of participants | 39.3 [32.0 to 47.0] | 43.8 [36.4 to 51.4] | 20.7 [14.9 to 27.5]
Statistical Analysis 1: Comparison: Asenapine 5 mg BID vs Placebo BID; Test type: Superiority or Other; p = 0.0001, Cochran-Mantel-Haenszel — Adjusted for region; Mean Difference (Final Values) = 18.6, 95% CI 2-sided [9.2 to 28.1] — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 2: Comparison: Asenapine 10 mg BID vs Placebo BID; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — Adjusted for region; Mean Difference (Final Values) = 23.1, 95% CI 2-sided [13.7 to 32.6] — Asenapine 10 mg BID minus Placebo BID

11. Secondary Outcome: Change From Baseline in Clinical Global Impressions -Severity of Illness (CGI-S) Score.
Description: The CGI-S is a score that measures the severity of overall bipolar illness. The score ranges on a scale from 1 to 7, where 1 is normal, and 7 is very severely ill. Change from baseline values that are negative represent an improvement in symptoms.
Time Frame: Baseline and Day 42
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Asenapine 5 mg BID | Asenapine 10 mg BID | Placebo BID
Number analyzed (Participants) | 173 | 178 | 174
Score on a scale | -0.69 [-0.86 to -0.52] | -0.77 [-0.94 to -0.61] | -0.18 [-0.35 to -0.01]
Statistical Analysis 1: Comparison: Asenapine 5 mg BID vs Placebo BID; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least square (LS) means difference = -0.52, 95% CI 2-sided [-0.75 to -0.28], Standard Error of Mean 0.12 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 2: Comparison: Asenapine 10 mg BID vs Placebo BID; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS mean difference = -0.59, 95% CI 2-sided [-0.82 to -0.36], Standard Error of Mean 0.12 — Asenapine 10 mg BID minus Placebo BID

12. Secondary Outcome: Percentage of Participants Who Were Clinical Global Impressions - Improvement (CGI-I) Responders.
Description: The CGI-I is a score on a 7-point scale for assessing the change from preceding phase of overall symptoms of bipolar disorder during the treatment of an acute episode or in longer term illness prophylaxis. Compared to the baseline, the CGI-I score ranges from 1 = very much improved since initiating treatment, to 7 = very much worse since initiating treatment. The CGI-I score was assessed at baseline and Day 42. Compared to the baseline measurement, a CGI-I responder had a score at Day 42 of 3 (minimally improved), 2 (much improved) or 1 (very much improved).
Time Frame: Day 42
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Asenapine 5 mg BID | Asenapine 10 mg BID | Placebo BID
Number analyzed (Participants) | 173 | 178 | 174
Percentage of participants | 63.6 [55.9 to 70.8] | 70.2 [62.9 to 76.8] | 41.4 [34.0 to 49.1]
Statistical Analysis 1: Comparison: Asenapine 5 mg BID vs Placebo BID; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — Adjusted for region; Mean Difference (Final Values) = 22.2, 95% CI 2-sided [12.0 to 32.4] — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 2: Comparison: Asenapine 10 mg BID vs Placebo BID; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — Adjusted for region; Mean Difference (Final Values) = 28.8, 95% CI 2-sided [18.9 to 38.8] — Asenapine 10 mg BID minus Placebo BID

ADVERSE EVENTS:
Time Frame: Up to 49 days for non-serious adverse events (AEs), and up to 79 days for serious AEs
Description: Participants who received at least one dose of trial medication
Arm/Group | Asenapine 5 mg BID | Asenapine 10 mg BID | Placebo BID
Serious Adverse Events (participants affected / at risk) | 10/175 | 5/181 | 13/174
Other Adverse Events (participants affected / at risk) | 96/175 | 110/181 | 89/174
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Asenapine 5 mg BID (N=175) | Asenapine 10 mg BID (N=181) | Placebo BID (N=174)
Sinus Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Subarachnoid Hemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Schizophrenia (Psychiatric disorders) | 8 (8) | 4 (4) | 8 (8)
Schizophrenia, paranoid type (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Asenapine 5 mg BID (N=175) | Asenapine 10 mg BID (N=181) | Placebo BID (N=174)
Constipation (Gastrointestinal disorders) | 10 (10) | 13 (15) | 11 (12)
Hypoaesthesia oral (Gastrointestinal disorders) | 19 (20) | 17 (18) | 6 (6)
Nasopharyngitis (Infections and infestations) | 13 (15) | 11 (13) | 8 (8)
Blood creatine phosphokinase increased (Investigations) | 3 (4) | 12 (12) | 4 (4)
Akathisia (Nervous system disorders) | 20 (22) | 19 (19) | 9 (9)
Dizziness (Nervous system disorders) | 7 (8) | 17 (17) | 5 (5)
Extrapyramidal disorder (Nervous system disorders) | 9 (9) | 14 (16) | 3 (3)
Headache (Nervous system disorders) | 11 (12) | 10 (12) | 11 (12)
Somnolence (Nervous system disorders) | 17 (17) | 22 (23) | 3 (3)
Insomnia (Psychiatric disorders) | 17 (18) | 14 (16) | 21 (23)
Schizophrenia (Psychiatric disorders) | 15 (15) | 25 (25) | 42 (44)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees to provide the sponsor 45 days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication that report any results of the trial. The sponsor shall have the right to review and comment with respect to publications, abstracts, slides, and manuscripts, and to review and comment on the data analysis and presentation.